CLINICAL TRIAL: NCT02405026
Title: HIV and Asthma in the Post-ART (Antiretroviral Therapy) Era
Brief Title: Determine the Prevalence and Severity of Asthma in HIV (Human Immunodeficiency Virus) Infected Patients
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00057348
Record Dates: First submitted 2014-12-15; First posted 2015-04-01 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Asthma; HIV
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, plasma, sputum supernatant, sputum cell pellet
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- HIV infected patients: HIV infected patients with asthma
- HIV uninfected patients: HIV uninfected patients with asthma
- HIV infected non-asthmatic patients: HIV infected patients without asthma

SUMMARY:
The purpose of this study is to determine the prevalence and severity of asthma in patients with HIV. To determine the immunological phenotype of HIV-infected patients with asthma.

DETAILED DESCRIPTION:
Prospectively clinically phenotype and the prevalence of asthma in HIV infected patients in the Duke ID Clinic

* HIV infected asthmatic subjects meeting clinical definitions for asthma compared to HIV uninfected asthma subjects identified at the DAAAC and HIV infected non-asthmatic subjects.
* Prospective immunological phenotyping - HIV-infected asthma subjects prospectively identified and clinically phenotyped compared to HIV-uninfected asthma subjects identified at the DAAAC and HIV infected non-asthma subjects.

Regarding the sampling method of probability sample: All samples for HIV infected asthmatic patients, HIV uninfected asthmatic patients and HIV infected non-asthmatics patients will be analyzed.

Retrospectively determine overall asthma prevalence and severity among HIV-infected patients. Retrospective immunological phenotyping (circulating cytokines) of HIV-infected patients utilizing available specimens in the Duke HIV Specimen Biorepository

* HIV-infected asthmatic subjects meeting asthma definition compared to overall asthma prevalence in U.S. population
* HIV-infected asthma subjects meeting asthma definitions compared to matched HIV-infected non-asthma subjects

ELIGIBILITY:
Inclusion Criteria:

* HIV infected asthmatic and non-asthmatic adults ≥18 years
* HIV uninfected asthma adults ≥18 years
* Females of childbearing potential have to be using medically acceptable contraceptive method for the duration of the study.
* Willing and able to give informed consent and adhere to visit/protocol schedules.
* Negative pregnancy test in women of childbearing potential
* For asthma patients: known or possible diagnosis of asthma for at least one year

Exclusion Criteria:

* Antibiotic administration for upper respiratory infection within the prior 30 days
* Greater than 10 pack a year smoking history
* No prior use of steroids (systemic) within the past 3 months
* Underlying illnesses that may result in altered lung function
* Students or employees who are under direct supervision of any Project or Core PI/Director.
* Pregnant or nursing mothers.
* Poorly controlled concomitant conditions as determined by the investigator.
* Subjects who have had an elective procedure (for example, colonoscopy, cystoscopy, etc.) within less than 2 weeks of the procedure date cannot be enrolled in the HIV Asthma study
* Subjects must delay enrollment by 2 weeks into the HIV Asthma study if they have received a single dose of systemic steroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV infected patients. Patients will be identified from the populations of the Duke Infectious Disease Clinic, and surrounding communities.
  HIV unifected patients. Patients will be identified through the Duke Asthma, Allergy and Airway Center, as well as from primary care physicians, and surrounding communities.
Sampling Method: Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2014-12; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Asthma prevalence of HIV infected subjects currently followed at the Duke Infectious Disease (ID) Clinic compared to HIV uninfected asthma subjects identified at the Duke Asthma, Allergy and Airway Center (DAAAC). | 12 months
  Assessed through Asthma control questionnaire, pulse oximetry, FeNO, Spirometry, Methacholine challenge, Induced sputum for differential, serum periostin, questionnaires
Asthma phenotypic characteristics of HIV infected subjects compared to HIV uninfected asthma subjects and HIV infected non-asthmatic subjects. | 12 months
  Assessed through blood collection

SECONDARY OUTCOMES:
Prospective immunological phenotyping of Th1/Th2/Th17 cytokines and T cell subsets | 12 months
  Assessed through blood sample collection
Retrospective immunological phenotyping (circulating cytokines) of HIV-infected patients utilizing available specimens in the Duke HIV Biorepository | 12 months
  The primary measure of is the quantitative difference in IL-6 between HIV-infected asthmatic subjects and HIV-infected non-asthmatic subjects.
Retrospectively determine overall asthma prevalence among HIV-infected patients | 12 months
  HIV-infected asthmatic subjects meeting electronic health records asthma definition Compared overall asthma prevalence in U.S. population.

CONTACTS AND LOCATIONS:
Overall Officials: Loretta Que, MD, Principal Investigator — Duke University
Locations (1):
- Duke Asthma Allergy and Airway Center, Durham, North Carolina, United States